CLINICAL TRIAL: NCT06237868
Title: The Effects of High-Frequency Repetitive Transcranial Magnetic Stimulation on Impulse Control Disorders in Parkinson's Disease Patients on Dopamine Replacement Therapy.
Brief Title: rTMS Over the Dorsolateral Prefrontal Cortex for the Treatment of Impulse Control Disorders in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Mariya V. Cherkasova, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2307823170
Record Dates: First submitted 2024-01-22; First posted 2024-02-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-04

CONDITIONS: Impulse Control Disorder; Parkinson Disease
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- rTMS Active (Active Comparator): the participant will receive a type of TMS called repetitive TMS (rTMS) wherein the magnetic pulses delivered will be close together in a rapid sequence over the dlPFC. Participants receive excitatory rTMS with a stimulation frequency of 20 Hz between 100-120% of their resting motor threshold.
  Interventions: Device: rTMS Active
- rTMS Sham (Sham Comparator): Sham rTMS will be the same as real rTMS, except a special sham coil will be used, which produces the same sensation on the scalp of the patients as the real coil but delivers no magnetic stimulation to the brain.
  Interventions: Device: rTMS Sham

INTERVENTIONS:
Device: rTMS Active — The participants undergo Active rTMS, approximately 10-15 min and then complete tasks and questionnaires.
  Arms: rTMS Active
Device: rTMS Sham — The participants undergo Sham rTMS, approximately 10-15 min and then complete tasks and questionnaires.
  Arms: rTMS Sham

SUMMARY:
This study's objective is to evaluate the effects of repetitive transcranial magnetic stimulation (rTMS) over the dorsolateral prefrontal cortex (dlPFC) of patients with Parkinson's Disease (PD) who experience impulse control disorders (ICDs) on impulse control symptoms and cognitive behaviors linked to ICDs: reinforcement learning and delay-discounting. This is a randomized sham-controlled cross-over trial. All patients will undergo a session of active rTMS and a session of sham rTMS, with the order of sessions randomized across participants. Following recruitment and eligibility screening, the eligible participants will undergo two sessions of rTMS (active and sham), immediately followed by neurocognitive tasks and questionnaires, no more than 1-2 weeks apart. Each session will have a duration of approximately 1-1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Clinician-confirmed diagnosis of PD
* Ability to provide informed consent, written and verbal
* Clinician-diagnosed impulse control disorder or impulse control behaviors including punding/hobbyism and dopamine dysregulation syndrome
* A Beck Depression Inventory (BDI) (Beck et al., 1961) score of 14 or lower
* A Montreal Cognitive Assessment (MoCA) (Nasreddine et al., 2005) score of 20 or higher
* On dopamine-replacement therapy

Exclusion Criteria:

* History of seizures or epilepsy
* History of brain lesions (such as multiple sclerosis, tumor) reported
* History of vascular issues in the brain, such as stroke
* History of a moderate to severe traumatic brain injury
* Meeting the criteria for a major psychiatric illness such as schizophrenia or depression (BDI score of 14 or higher).
* Having significant cognitive impairment (assessed by MoCA, cutoff score of 20) (Nasreddine, et al., 2005)
* Having had TMS done in the recent past (within a year)
* Pregnancy assessed in female patients
* Intracranial metallic objects (except for dental fillings)
* Current use of substances or medications known to significantly reduce seizure threshold.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Delay-Discounting | Baseline to 1 hour following the intervention
  Change in performance on a task assessing delay-discounting. Delay-discounting assesses the participants' impulsivity by requiring them to make choices between smaller sooner hypothetical money rewards and larger later hypothetical money rewards (e.g. $10 today vs $100 in a year). This is a hypothetical choice, and the participant will not be receiving the chosen rewards. A short preliminary version of the task will be completed at the start of the first session (prior to TMS) to optimize task parameters for each participant. The task will be completed on a laptop computer.
Change in Reinforcement Learning | Baseline to 1 hour following the intervention
  Change in performance on a task assessing reinforcement learning. The reinforcement learning task assesses how well participants learn from rewards vs. punishments. The task will ask participants to choose from two stimuli that predict reward (gaining points) or punishment (losing points) at different rates, which they will learn in the course of the task based on feedback. At the end of the task, participants will be asked to rate how well each stimulus predicted reward or punishment.

SECONDARY OUTCOMES:
Change in impulse control disorder symptoms | Baseline to 1 hour following the intervention
  Change in impulse control disorder symptoms measured using a modified version of the Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS). QUIP-RS is a self-administered assessment of impulsive and compulsive behaviors in patients with PD. The QUIP-RS is a brief 28-item patient-reported or clinician-rated scale that was developed in PD and derived from the QUIP to measure of severity of ICDs. Each item is rated on a 5-point Likert scale assessing the frequency of symptoms with a range of scores from 0 (never) to 4 (very often).

CONTACTS AND LOCATIONS:
Overall Officials: Mariya V Cherkasova, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No